CLINICAL TRIAL: NCT05320536
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Clinical Study of Gulingji Capsule in the Treatment of Idiopathic Oligospermia, Asthenia, and Teratozoospermia.
Brief Title: A Clinical Study of Gulingji Capsule in the Treatment of Idiopathic Oligospermia, Asthenia, and Teratozoospermia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Reproductive Medicine Center, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guilingji Capsule treatment
Record Dates: First submitted 2021-12-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia | interventions — guilingji

STUDY DESIGN:
Intervention Model Description: Blind-wrapped drugs and corresponding emergency envelopes will be distributed to each centre in serial numbers based on the number of patients assigned to each centre. Each center shall sign a drug acceptance form, signed by two people in duplicate, with the group leader and each center holding one copy. The experimental drugs are stored at room temperature, away from light and dry, and are in the charge of special personnel. Each center will distribute drugs to eligible patients starting with the minimum number.
Who Masked: Participant, Investigator
Masking Description: The group randomization method was adopted according to the central stratification, and a total of 240 cases were randomly assigned equally to the experimental group and the control group by SAS 9.2 statistical system programming to generate a random allocation sequence table. Sequence table according to the distribution of drugs for blind packaging, medicine make blind by the personnel not to participate in clinical trials according to the generated random distribution plans and standard operating procedures for blind of experimental drugs allocation coding, coding procedure shall monitor, after completion of blind plait blind bottom seal should be in duplicate, respectively by the eastern theatre, head of the general hospital drug clinical trial institution and subject to save. SAS programs that generate randomization and related parameters are saved together with the blind end.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Guilingji capsule Take 2 tablets orally, once before breakfast and dinner, and take them with saline. The total treatment period is 90 days.
  Interventions: Drug: Guilingji Capsule
- Control group (Placebo Comparator): Placebo Take 2 tablets orally, once before breakfast and dinner, and take them with saline. The total treatment period is 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guilingji Capsule — This medicine is capsule medicine, take method is oral.
  Arms: Experimental group
Drug: Placebo — This medicine is capsule medicine（Placebo）, take method is oral.
  Arms: Control group

SUMMARY:
The object of study for patients with idiopathic disease of OAT, the use of multicenter, randomized, double-blind, controlled, prospective clinical research, choose according to row, standard units of idiopathic male infertility clinics less weak abnormal sperm, randomly divided into experimental group and the placebo group, the comparison between the two groups of patients and semen parameters before and after medication, seminal plasma hormone, serum lipid levels and other indicators;At the same time, serum and seminal plasma samples of the two groups of patients before and after treatment were collected for bioinformatics analysis of protein spectrum to find the effector molecules of Gulingji capsule.

DETAILED DESCRIPTION:
The WHO defines infertility as a condition in which a couple cohabitates and has normal sex, has not used contraception for more than a year and the woman has not been able to conceive naturally.Some male infertility patients who cannot find related infertility factors are called idiopathic male infertility.These male infertility patients are often characterized by abnormal sperm count (including oligospermia, azoospermia, occult sperm), abnormal motility (including asthenospermia, asthenospermia), or malformed sperm, collectively referred to as idiopathic oligospermia (idiopathic OAT).

At present, the treatment methods of idiopathic OAT are mostly empirical treatment, including anti-oxidation treatment, treatment to improve cell energy metabolism, treatment to improve microcirculation of the whole body and reproductive system, etc.In general, traditional Chinese treatment should be combined with traditional Chinese medicine.However, the relevant mechanism of TCM treatment of OAT is not yet clear.

The object of study for patients with idiopathic disease of OAT, the use of multicenter, randomized, double-blind, controlled, prospective clinical research, choose according to row, standard units of idiopathic male infertility clinics less weak abnormal sperm, randomly divided into experimental group and the placebo group, the comparison between the two groups of patients and semen parameters before and after medication, seminal plasma hormone, serum lipid levels and other indicators;At the same time, serum and seminal plasma samples of the two groups of patients before and after treatment were collected for bioinformatics analysis of protein spectrum to find the effector molecules of Gulingji capsule.

It is assumed that the probable case loss rate in the trial is 20%, with 120 cases in each group, and a total of 240 cases are required.

Drug treatment: Gulingji capsule was taken orally for 2 capsules, once before breakfast and dinner, and was taken with saline solution. The total treatment period was 90 days.(Placebo is rice flour)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as oligoasthenospermia according to the World Health Organization Laboratory Manual for Human Semen Examination and Treatment (5th edition);
2. initial examination and reexamination of abnormal semen quality shall meet one of the following conditions: sperm density < 15×10^6 / mL or total sperm count < 39×10^6, proportion of forward motile sperm < 32% or total sperm viability < 40%, percentage of normal sperm < 4%.

Exclusion Criteria:

1. Leucospermia, with testis, epididymitis, prostatitis, severe genital trauma, testicular torsion, urinary tract infection, cryptorchidism, varicocele, and a history of serious medical conditions such as diabetes, tumor history, inguinal and genital surgery.
2. Testicular volume < 12ml (B-ultrasonic measurement).
3. BMI < 18.5 or > 32.
4. Chromosomal karyotype abnormalities.
5. Patients with endocrine diseases.
6. Exposure to an occupation or environment with reproductive toxicity.
7. Drug therapy to improve semen quality has been used in the past 2 weeks.
8. Hepatobiliary disease, severe renal insufficiency, clinical disease or history of medication known to reduce fertility.
9. A known or suspected history of allergy to experimental drugs and similar products.
10. Any circumstance that the investigator considers to be likely to interfere with participation in the study or assessment.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
TNPMS | 1 years
  Total sperm count in forward motion

SECONDARY OUTCOMES:
DFI | 1 years
  Sperm DNA fragmentation rate

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Center for Reproductive Medicine, Jinling Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Jiangsu
  - Xi 'an Tangdu Hospital, Xi’an, Jiangsu

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05320536/Prot_SAP_ICF_000.pdf